CLINICAL TRIAL: NCT07144761
Title: Evaluating Patient Reported Outcomes and Surgeon Satisfaction With Ziplyft™
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Osheru Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 6520-Osheru
Record Dates: First submitted 2025-06-16; First posted 2025-08-27 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Blepharoplasty

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Ziplyft Device (Experimental): Ziplyft is a Class 1, 510(k) Exempt device for removing excess unwanted eyelid skin.
  Interventions: Device: Ziplyft

INTERVENTIONS:
Device: Ziplyft — Ziplyft™ is a Class 1, 510(k) Exempt device for removing excess unwanted eyelid skin using a novel surgical device called Ziplyft™.

SUMMARY:
The objective of this study is to evaluate patient-reported outcomes, surgeon reported outcomes, bruising, symmetry, the success of tissue adhesive for wound closure, and case time.

ELIGIBILITY:
Inclusion Criteria:

1. Provide signed written consent prior to participation in any study-related procedures.
2. Ability, comprehension, and willingness to follow study instructions, and likely to complete all study visits.
3. Male or female adults, ≥ 35 years old at the Preoperative Visit
4. Willing to return for required follow-up visits.
5. Subjects with excess eyelid skin are eligible to undergo the procedure in the opinion of the investigator.
6. Female subjects must be 1-year postmenopausal, surgically sterilized, or, if of childbearing potential, have a negative urine pregnancy test at the Preoperative Visit. Women of childbearing potential must use an acceptable form of contraception throughout the study. Acceptable methods include at least one of the following: intrauterine (intrauterine device), hormonal (oral, injection, patch, implant, ring), barrier with spermicide (condom, diaphragm), or abstinence.

Exclusion Criteria:

1. Subjects with a current Ptosis diagnosis
2. Subjects with a history of Graves' Disease
3. Subjects with Myasthenia Gravis
4. Subjects that in the opinion of the investigator are anatomically not conducive to using devices (e.g., heavy brow, severe hollowing of the upper eyelid, history of ocular or orbital trauma).
5. Subjects that have had any previous surgery eyelid or eyebrow region.
6. Use of anticoagulation therapy, including, but not limited to Aspirin, NSAIDS, Ibuprofen within 7 days and Xarelto, Warfarin, Enoxaparin, Plavix within 3 days prior to planned study procedure.
7. Active or recent (within 3 months) tobacco user
8. Allergy to adhesive glue
9. Participation in any study of an investigational, interventional product within 30 days prior to the Preoperative Visit or at any time during the study period.
10. Pregnant or nursing females.

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Improvement in overall patient satisfaction - Satisfaction with facial appearance and eyes | From enrollment to the last visit at 3 months
  Demonstrate an improvement in overall patient satisfaction by comparing pre-operative and post-operative patient reported outcome scores.
  FACE-Q - Aesthetics - Appearance - Satisfaction with facial appearance FACE-Q - Aesthetics - Appearance - Satisfaction with Eyes
  On a scale of 1-4 Very Dissatisfied being 1 and Very Satisfied being 4
Surgeon Satisfaction and Efficiency | From enrollment to the last visit at 3 months.
  Demonstrate surgeon satisfaction and efficiency with Ziplyft™, measured by Surgeon Satisfaction Survey with questions focused on ease of procedure, patient tolerance, device useability, surgical technique, procedural time, wound closure, need for suture, ease of achieving symmetry, device placement on the lid crease, cutting mechanism, seal of the zipper-locked tissue, surgical time and evaluating for post-operative complications with 5 being better outcome and 1 being worse.
Improvement in Eye Age | From enrollment to the last visit at 3 months.
  Demonstrate improvement in Eye Age and Face Age after the Ziplyft™ procedure.
  FACE-Q - Aesthetics - Appearance - Aging Appraisal On a scale of 1-4, with 1 being Definitely Disagree and 4 being Definitely agree
Measure the success of tissue adhesive for wound closure. | From enrollment to the last visit at 3 months.
  Measuring the success of the tissue adhesive involves evaluating the following: Visual inspection, Adhesion strength and adherence, and Patient satisfaction. Questions added in the patient satisfaction survey about comfort of glue, ease of blinking, aesthetically acceptable with 1 being a worse outcome and 4 being better.
Post-operative ecchymosis | From enrollment to the last visit at 3 months.
  Document post-operative ecchymosis with Ziplyft. Measured by post-operative photographs.
Eyelid Symmetry | From enrollment to the last visit at 3 months.
  To achieve optimal eyelid symmetry after eyelid surgery with Ziplyft™ by independent reviewers' assessments.
  Measurement of symmetry will be judged on a scale of 1-4 by an independent reviewer based on post-op patient photos. 1 being worse and 4 being better outcome.
Improved case time | From enrollment to last visit at 3 months.
  Demonstrate improved case time with Ziplyft™

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Center for Excellence in Eye Care, Miami, Florida
  - Vance Thompson Vision, Alexandria, Minnesota
  - Eye Care Specialists, Kingston, Pennsylvania
  - Vance Thompson Vision, Sioux Falls, South Dakota
  - The Eye Centers of Racine and Kenosha, LTD, Kenosha, Wisconsin

IPD SHARING:
Plan to Share IPD: No